CLINICAL TRIAL: NCT05426382
Title: Sidekick Health Digital Solution (SK-241) for Individuals With Non Alcoholic Fatty Liver Disease (NAFLD): A Feasibility Study
Brief Title: A Digital Solution for Individuals With Non Alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidekick Health (Industry)
Collaborators: Hjartamiðstöðin, Iceland (Unknown); Hjartavernd, Iceland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SK-241-NAFLD
Record Dates: First submitted 2022-06-10; First posted 2022-06-22 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: non alcoholic fatty liver disease; digital solution; lifestyle change; remote monitoring; clinical outcome; quality of life; digital intervention; non-alcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Multi-center single-arm open label intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital solution group (Experimental): Participants will be instructed to download a lifestyle-changing mobile application to which they will have access for 9 months. The program aims to provide remote symptom monitoring by a health coach and by having participants enter data (on diet, exercise, weight, stress and energy levels, etc) and patient reported outcomes (PROs) via the SidekickHealth platform to empower positive lifestyle changes.
  The intervention consists of a 12-week digital behavioral change program with an additional 6-month maintenance program, during which time the patient still has access to the application but with limited features compared to the first 12 weeks. During the total 9-month study period all participants will also receive standard of care.
  Interventions: Device: A digital care solution for patients with NAFLD

INTERVENTIONS:
Device: A digital care solution for patients with NAFLD — A digital solution that provides remote symptom monitoring and support of healthy lifestyle choices through tasks that are made more attractive with gamification and rewards.
  Other Names: SK-241

SUMMARY:
Sidekick Health has developed a digital behavioral change program (SK-241) specifically designed for people with metabolic derangements and non-alcoholic fatty liver disease (NAFLD). The SK-241 is delivered through a mobile application and aims at improving lifestyle and health outcomes by focusing on improving diet, increasing activity levels and reducing stress. In this study, the feasibility of the newly developed digital behavioral change program (SK-241) will be evaluated in a minimum of 30 individuals with a NAFLD diagnosis. The primary aim is to explore the acceptability of the SK-241 program by its users, in addition to exploring changes in clinical outcomes and medication adherence after a 12-week intervention with 6 months follow up.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is an umbrella term used to describe a spectrum of liver pathology, characterized by >5% fat accumulation in the liver (steatosis), among people who drink little or no alcohol. Both genetic and lifestyle-related factors contribute to the pathogenesis of NAFLD. It is strongly associated with metabolic derangements, obesity, insulin resistance and type 2 diabetes mellitus. NAFLD is considered the liver manifestation of metabolic syndrome.

NAFLD can progress from a simple steatosis to a more severe and progressive condition, referred to as non-alcoholic steatohepatitis (NASH), which is characterized by additional liver inflammation and hepatocyte injury with or without fibrosis. In general, 20% of NAFLD patients are believed to progress to NASH.

Finding convenient and effective ways to incorporate lifestyle changes into daily lives of people with NAFLD and NASH is important. Sidekick Health has developed a digital behavioral change program (SK-241) for NAFLD and NASH patients consisting of an interactive mobile application.

The aim of this study is primarily to assess the acceptability and feasibility of adding a digital lifestyle intervention (SK-241) to the standard of care (SoC) for NAFLD patients, by assessing participants engagement, retention and satisfaction with the SK-241 program in a minimum of 30 individuals with a NAFLD diagnosis. In addition, the clinical effectiveness of the program will be explored. A minimum of 30 individuals with a NAFLD diagnosis will be included for a 12-week intervention with 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a NAFLD diagnosis, defined as:

Confirmed liver steatosis >5%, with a FibroScan CAP cutoff score of > 294 decibel (dB)/m among individuals with one or more of the following: Type 2 diabetes OR BMI>30 OR Metabolic syndrome OR Previous diagnosis of NAFLD within the last 12 months

* for individuals with type 2 diabetes: Stable dose of antidiabetic medication the last 90 days before screening (metformin, glitazones, glucagon like peptide-1 (GLP-1) analogues, sodium-glucose co transporter-2 (SGLT-2) inhibitor, sulfonylurea, insulin)
* Capacity to give informed consent and understands verbal and written Icelandic
* Owns and knows how to operate a smartphone
* Willing and able to comply with the study intervention, all scheduled visits and procedures

Exclusion Criteria:

* Insulin use
* Known or self-reported cirrhosis
* Alcohol consumption over 14 units/week for males, 7 units/week for women
* Self-reported Hepatitis B (HepB), Hepatitis C (HepC), human immunodeficiency virus (HIV), or autoimmune hepatitis
* Vitamin E intake of > 400 IU/day - unless stable for 12 weeks prior to baseline
* Taking medications associated with liver steatosis; steroids, methotrexate, tamoxifen, amiodarone, tetracycline, valproic acid
* Self-reported pregnancy
* Participation in a weight loss program
* History of, or any existing medical condition (e.g., ongoing cancer treatment, severe cardiopulmonary- or musculoskeletal disease, stroke, or myocardial infarction in the last 6 months) that, in the opinion of the investigator, would interfere with evaluation of the study intervention or affect the interpretation of the results of the study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Acceptability and feasibility of the digital program (SK-241) - retention. | 12 weeks
  Assess retention by percentage of users that complete the SK-241 program at week 12. 'Complete the program' is defined as finishing 75% of the program.
Acceptability and feasibility of the digital program (SK-241) - engagement. | 12 weeks
  Assess engagement by percentage of users that are active in the SK-241 program during the 12 weeks. 'Active' is defined as visiting the application at least once per week.
Acceptability and feasibility of the digital program (SK-241) - satisfaction. | 12 weeks
  Assess satisfaction based on the scores in the 18-item mobile health (mHealth) App Usability Questionnaire at week 12.
  Answers are scored on a 7-point Likert scale (ranging from 1 for "strongly disagree"to 7 "strongly agree") and total scores range from 18 to 126. The higher the score, the better the usability.

SECONDARY OUTCOMES:
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on weightloss. | 9 months
  Change in weight, from baseline to week 12 and month 9
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on HbA1c. | 9 months
  Changes, from baseline to week 12 and month 9 in:
  Hemoglobin A1c (HbA1c), expressed in millimol per mol (mmol/mol).
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on fasting glucose. | 9 months
  Changes, from baseline to week 12 and month 9 in:
  fasting glucose, measured in millimol per liter (mmol/L)
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on fasting insulin. | 9 months
  Changes, from baseline to week 12 and month 9 in:
  fasting insulin, measured in picomol per liter (pmol//L)
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on liver function. | 9 months
  Changes, from baseline to week 12 and month 9, in liver enzymes in the serum:
  Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Gamma- Glutamyl Transferase (GGT), all measured in international units per liter (IU/L)
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on cholesterol. | 9 months
  Changes, from baseline to week 12 and month 9 in:
  Total cholesterol, Low Density Lipoprotein - Cholesterol (LDL-C), High Density Lipoprotein - Cholesterol (HDL-C), and triglycerides. These are all measured in millimol per liter (mmol/L)
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on hs-CRP. | 9 months
  Changes, from baseline to week 12 and month 9, in:
  high-sensitivity C-reactive protein (hs-CRP), measured in milligram per liter (mg/L)
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on the cardiovascular risk factor blood pressure | 9 months
  Changes, from baseline to week 12 and month 9, in:
  Blood pressure in millimeters of mercury (mmHg)
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on the cardiovascular risk factor waist circumference. | 9 months
  Changes, from baseline to week 12 and month 9, in:
  Waist circumference in centimeters (cm)
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on the cardiovascular risk factor activity level. | 9 months
  Changes, from baseline to week 12 and month 9, in:
  Activity level, as assessed with an in-app step counter, and measured in number of steps
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on body composition. | 9 months
  Changes in body composition (fat mass and lean mass), measured by dual-energy X-ray absorptiometry (DXA) at baseline, week 12 and 9 months.
  Fat mass and lean mass are both expressed as percentage (%).
The feasibility of adding a digital program (SK-241) to standard of care, by exploring its effects on liver fat content. | 9 months
  Changes in liver fat fraction (%) assessed by magnetic resonance imaging-proton density fat fraction (MRI-PDFF) at baseline, week 12 and 9 months.
The feasibility of adding a digital program (SK-241) to standard of care, by assessing health related quality of life (HRQoL) | 9 months
  Changes in self-reported scores on the EuroQuol Five Dimension - Five Level (EQ-5D-5L) health questionnaire from baseline to week 12 and month 9.
  EQ-E5-5L scores range from -0.530 to 1, with higher scores indicating a better health status. A score of 1 indicates full health.
The feasibility of adding a digital program (SK-241) to standard of care, by assessing mental health. | 9 months
  Changes in self-reported scores of the Depression, Anxiety and Stress Scale - 21 Items (DASS-21) questionnaire from baseline to week 12 and month 9.
  Each question has a Likert scale of 4 options where 0 represents "did not apply to me" to 3 "applied to me very much". The scores on the subscales range from 0 to 42, and low scores indicate a better mental health status.
The feasibility of adding a digital program (SK-241) to standard of care, by assessing medication adherence. | 9 months
  Changes in self-reported scores on the Morisky Medication adherence Scale (MMAS-8) questionnaire from baseline to week 12 and month 9. The MMAS-8 is an 8-item structured, self-reported medication adherenece measure.
  Scores on the MMAS-8 range from 0-8, with 0 reflecting high adherence, 1-2 medium adherence and 3-8 low adherence.

OTHER OUTCOMES:
Exploratory objective: liver steatosis | 9 months
  Changes in Controlled Attenuation Parameter (CAP) Fibroscan score. CAP Fibroscan score is measured in decibels per meter (dB/m) and assessed at baseline, week 12 and 9 months.
  CAP Fibroscan scores range from from 100 to 400 dB/m, with a lower score indicating a better outcome as it indicates less liver steatosis.
Exploratory objective: liver fibrosis | 9 months
  Changes in Liver Stiffness Measurement (LSM) Fibroscan score.The LSM Fibroscan scores are measured in kilopascal (kPa) and assessed at baseline, week 12 and 9 months.
  LSM FibroScan scores range from 2.5 kPa to 75 kPa. A lower scores indicates a better outcome.
Safety objective: Monitor the safety and any potential adverse effects of the digital solution on patients and outcomes. | 9 months
  Incidence of adverse events (AE) and serious adverse events (SAE) reportings at week 12 and 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sigríður Björnsdóttir, MD PhD, Principal Investigator — Hjartamiðstöðin
Locations (2):
- Iceland (2):
  - Hjartamiðstöðin, Kopavogur
  - Hjartavernd, Kopavogur

IPD SHARING:
Plan to Share IPD: No
Anonymized Individual Participant Data (IPD) may be shared with other researchers for relevant research purposes following complementary ethical review and approval from the Ethical Review Board.

REFERENCES:
- [Derived] Bjornsdottir S, Ulfsdottir H, Gudmundsson EF, Sveinsdottir K, Isberg AP, Dobies B, Akerlie Magnusdottir GE, Gunnarsdottir T, Karlsdottir T, Bjornsdottir G, Sigurdsson S, Oddsson S, Gudnason V. User Engagement, Acceptability, and Clinical Markers in a Digital Health Program for Nonalcoholic Fatty Liver Disease: Prospective, Single-Arm Feasibility Study. JMIR Cardio. 2024 Feb 15;8:e52576. doi: 10.2196/52576. PMID 38152892